CLINICAL TRIAL: NCT06649656
Title: A Multicenter, Open Label Phase I Clinical Trial Evaluating the Safety and Pharmacokinetics of TQB2252 Injection in Subjects With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2252-I-01
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-06

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2252 injection (Experimental): This product is administered via intravenous infusion, with recommended doses of 600mg TQB2223 monoclonal antibody and 200mg penpulimab injection, administered once every 3 weeks.
  Interventions: Drug: TQB2252 injection

INTERVENTIONS:
Drug: TQB2252 injection — TQB2252 injection is a compound preparation of TQB2223 monoclonal antibody (LAG-3) and penpulimab (PD-1), with a specification of 300mg TQB2223 monoclonal antibody and 100mg (20ml) penpulimab per bottle.

SUMMARY:
This study is a multicenter, single arm, and open design Phase I clinical trial aimed at evaluating the safety, Pharmacokinetics (PK) characteristics, immunogenicity, and preliminary efficacy of TQB2252 injection in subjects with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study, signed an informed consent form, and showed good compliance;
* 18 years old ≤ 75 years old (calculated from the date of signing the informed consent form);
* Electrocorticogram (ECOG) score ranges from 0 to 1 points;
* Expected survival is greater than 12 weeks；
* Confirmed to have at least one measurable lesion according to RECIST 1.1 (solid tumor) or Lugano 2014 (lymphoma) criteria；
* Late stage malignant tumor subjects who have failed standard treatment or lack effective treatment；
* Women of childbearing age should agree to use effective contraceptive measures during the study period and for 6 months after the end of the study; Men should agree to use effective contraceptive measures during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Has experienced or currently has other malignant tumors within the past 5 years prior to the first use of medication;
* There are multiple factors that affect diseases related to intravenous injection and venous blood collection;
* The adverse reactions of previous anti-tumor treatments have not recovered to a Common Terminology Criteria for Adverse Events (CTCAE) v5.0 score of ≤ 1;
* Individuals who have undergone major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the expected study treatment period within 4 weeks prior to the first use of medication;
* Subjects who experience any bleeding or bleeding events ≥ CTCAE grade 3 within 4 weeks prior to the first administration;
* An arterial/venous thrombotic event occurred within 6 months prior to the first administration;
* Active viral hepatitis with poor control;
* Active syphilis infected individuals in need of treatment;
* History of active pulmonary tuberculosis, idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or clinically symptomatic active pneumonia;
* Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
* Diagnosed with immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy due to a history of hepatic encephalopathy;
* Previously experienced grade 3 or higher adverse reactions related to immunotherapy;
* Suffering from significant cardiovascular disease;
* Active or uncontrolled severe infections;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases;
* Individuals with epilepsy who require treatment;
* Previously received treatment with similar anti-lag3 drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) rate | From date of the first dose until the date of 28 days after last dose or new anti-tumor treatment, whichever came first.
  The evaluation criteria for the nature and severity of adverse events are based on the National Cancer Institute's CommonTerminology Criteria for Adverse Events (NCI CTCAE version 5.0).

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (Tmax) | Day1 of Cycle1, Cycle3: within 30 minutes pre-dose, 0.25, 2, 4, 8, 24, 48, 168, 336 hour post dose. Day1 of Cycle2, Cycle4～Cycle 8: pre-dose. (Each cycle is 21 days)
  Time to reach maximum (peak) plasma concentration following drug administration
Maximum Plasma Concentration (Cmax) | Day1 of Cycle1, Cycle3: within 30 minutes pre-dose, 0.25, 2, 4, 8, 24, 48, 168, 336 hour post dose. Day1 of Cycle2, Cycle4～Cycle 8: pre-dose. (Each cycle is 21 days)
  The Cmax is the maximum observed plasma concentration of TQB2252.
Elimination half-life (t1/2) | Day1 of Cycle1, Cycle3: within 30 minutes pre-dose, 0.25, 2, 4, 8, 24, 48, 168, 336 hour post dose. Day1 of Cycle2, Cycle4～Cycle 8: pre-dose. (Each cycle is 21 days)
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Objective Response Rate (ORR) | up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
Progression-free survival (PFS) | up to 2 years
  Defined as the time from the first dose of TQB2252 to the first occurrence of disease progression or death from any cause.
Disease control rate (DCR) | up to 2 years
  Defined as the proportion of subjects with CR, PR, or Stable Disease (SD).
Duration of Response (DOR) | up to 2 years
  Defined as the time from first documented response to documented disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China